CLINICAL TRIAL: NCT01823835
Title: An Open-Label, Phase Ia/Ib/IIa Study of GDC-0810 Single Agent or in Combination With Palbociclib and/or an LHRH Agonist in Women With Locally Advanced or Metastatic Estrogen Receptor Positive Breast Cancer
Brief Title: A Study of GDC-0810 Single Agent or in Combination With Palbociclib and/or a Luteinizing Hormone-Releasing Hormone (LHRH) Agonist in Women With Locally Advanced or Metastatic Estrogen Receptor Positive Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to halt the development of GDC-0810, but not due to any safety concerns.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29642; 2014-004852-77 (EudraCT Number)
Record Dates: First submitted 2013-03-25; First posted 2013-04-04 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 3-(4-(2-(2-chloro-4-fluorophenyl)-1-(1H-indazol-5-yl)but-1-en-1-yl)phenyl)acrylic acid; Gonadotropin-Releasing Hormone; palbociclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Phase Ia - Cohort 1 (Experimental): 100 mg GDC-0810 once daily (QD) in fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 2 (Experimental): 200 mg GDC-0810 QD in fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 3 (Experimental): 400 mg GDC-0810 QD in fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 4 (Experimental): 600 mg GDC-0810 QD in fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 5 (Experimental): 600 mg GDC-0810 QD in non-fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 6 (Experimental): 300 mg GDC-0810 twice daily (BID) in fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 7 (Experimental): 800 mg GDC-0810 QD in fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 8 (Experimental): 800 mg GDC-0810 QD in non-fasting state.
  Interventions: Drug: GDC-0810
- Phase Ia - Cohort 9 (Experimental): 400 mg GDC-0810 BID in fasting state.
  Interventions: Drug: GDC-0810
- Phase IIa - Cohort A1 (Experimental): 600 mg GDC-0810 QD. Additionally, participants in this arm did not receive any prior treatment with fulvestrant and had confirmed ER-a (ESR1) mutation of the ligand binding domain (LBD).
  Interventions: Drug: GDC-0810
- Phase IIa - Cohort A2 (Experimental): 600 mg GDC-0810 QD. Additionally, participants in this arm had prior treatment with fulvestrant and confirmed ER-a (ESR1) mutation of the LBD.
  Interventions: Drug: GDC-0810
- Phase IIa - Cohort B1 (Experimental): 600 mg GDC-0810 QD. Additionally, participants in this arm did not receive any prior treatment with fulvestrant and had progressed following ≤1 prior therapy with an aromatase inhibitor (AI).
  Interventions: Drug: GDC-0810
- Phase IIa - Cohort B2 (Experimental): 600 mg GDC-0810 QD. Additionally, participants in this arm had prior treatment with fulvestrant and progressed following ≤1 prior therapy with an AI.
  Interventions: Drug: GDC-0810
- Phase Ib - Cohort C1 (Experimental): 400 mg GDC-0810 + 125 mg Palbociclib QD.
  Interventions: Drug: GDC-0810; Drug: Palbociclib
- Phase Ib - Cohort D1 (Experimental): ≤600 mg GDC-0810 QD + LHRH agonist once monthly.
  Interventions: Drug: GDC-0810; Drug: LHRH Agonist

INTERVENTIONS:
Drug: GDC-0810 — GDC-0810 administered orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, GDC-0810 drug supply exhausted, or study termination (up to 3 years).
Drug: LHRH Agonist — LHRH agonist administered once monthly until disease progression, unacceptable toxicity, withdrawal of consent, GDC-0810 drug supply exhausted, or study termination (up to 3 years). Choice of LHRH agonist will be an institutional choice approved for use in breast cancer.
  Arms: Phase Ib - Cohort D1
Drug: Palbociclib — Palbociclib administered orally once daily until disease progression, unacceptable toxicity, withdrawal of consent, GDC-0810 drug supply exhausted, or study termination (up to 3 years).
  Arms: Phase Ib - Cohort C1

SUMMARY:
This study is a multi-institution, Phase Ia/Ib/IIa open-label, dose-finding, safety, pharmacokinetics (PK), and proof-of-concept study of GDC-0810 as a single agent and in combination with palbociclib and/or LHRH agonist. The study is divided into 3 phases: Phase Ia, Phase Ib, and Phase IIa. During Phase Ia (dose escalation phase), GDC-0810 single agent will be administered orally on a continuous daily dosing regimen with a Day -7 lead-in period for single dose PK evaluation prior to the start of daily treatment. The incidence of dose-limiting toxicities (DLTs) will be evaluated from Day -7 through the first cycle (28 days) of treatment (35 days total). Depending on safety and tolerability, participants will be assigned sequentially to escalating doses of GDC-0810 using standard 3 + 3 design. During Phase Ib (dose escalation and expansion phase), participants will receive GDC-0810 with palbociclib and/or LHRH agonist to determine the recommended Phase II dose (RP2D) and assess the safety and tolerability of concomitant administration. During Phase IIa (dose expansion phase), participants previously treated with an aromatase inhibitor (AI) will be treated at the RP2D to further characterize the safety, PK, pharmacodynamics, and anti-tumor activity of GDC-0810.

ELIGIBILITY:
Inclusion Criteria:

Phase 1a portion

* Histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of either locally recurrent disease not amenable to resection or radiation therapy with curative intent, or metastatic disease, both progressing after at least 6 months of hormonal therapy for estrogen receptor (ER) positive breast cancer
* ER-positive, human epidermal growth factor 2 (HER2) negative
* At least 2 months must have elapsed from the use of tamoxifen
* At least 6 months must have elapsed from the use of fulvestrant
* At least 2 weeks must have elapsed from the use of any other anticancer hormonal therapy
* At least 3 weeks must have elapsed from the use of any chemotherapy
* Postmenopausal status
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate organ function

Phase Ib portion

* All above inclusion criteria, except:
* Postmenopausal status, pre- and peri-menopausal participants will also be included
* ECOG performance status less than 2
* At least 2 months must have elapsed from the use of tamoxifen not applicable
* At least 6 months must have elapsed from the use of fulvestrant not applicable

and plus:

* Documented sensitivity to prior hormonal therapy
* Cohort C1 (palbociclib combination cohorts): no prior treatment with cyclin-dependent kinase (CDK) 4/6 inhibitor

Phase IIa portion

* All above inclusion criteria for Phase Ia, except:
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* At least 6 months must have elapsed from the use of fulvestrant not applicable

and plus:

* Cohort A only: confirmed estrogen receptor alpha (ESR1) mutation and presence of measurable disease as per RECIST v1.1 or evaluable bone disease
* Cohort A1 only: no prior fulvestrant allowed; at least 2 months must have elapsed from the use of tamoxifen
* Cohort A2 only: prior fulvestrant allowed
* Cohort B only: disease progression following no more than 1 prior treatment with an aromatase inhibitor in the advanced/metastatic setting
* Cohort B1 only: no prior fulvestrant allowed
* Cohort B2 only: prior fulvestrant allowed

Exclusion Criteria:

Phase 1a portion

* Untreated or symptomatic central nervous system (CNS) metastases
* Endometrial disorders
* More than 2 prior chemotherapy in the advanced/metastatic setting (prior adjuvant chemotherapy is allowed so long as it occurred greater than or equal to 12 months prior to enrollment)
* Current treatment with any systemic anticancer therapies for advanced disease
* Any significant cardiac dysfunction within 12 months prior to enrollment
* Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or upper gastrointestinal surgery including gastric resection
* Known human immunodeficiency virus (HIV) infection
* Known clinically significant history of liver disease
* Major surgery within 4 weeks prior to enrollment
* Radiation therapy within 2 weeks prior to enrollment

Phase Ib portion - all above exclusion criteria, plus:

* Cohort C1 (palbociclib combination cohorts): history of venous thromboembolic event requiring therapeutic anticoagulation; vaginal bleeding within 2 months prior to enrollment

Phase IIa portion - all above exclusion criteria, plus:

* Cohort A1, A2, and Cohort B2 only: more than 1 prior chemotherapy in the advanced/metastatic setting
* Cohort B1 only: prior chemotherapy in the advanced/metastatic setting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (8):
  - Ucsd Medical Center, San Diego, California
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Mount SInai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- VU MEDISCH CENTRUM; Dept. of Medical Oncology, Amsterdam, Netherlands
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Bardia A, Mayer I, Winer E, Linden HM, Ma CX, Parker BA, Bellet M, Arteaga CL, Cheeti S, Gates M, Chang CW, Fredrickson J, Spoerke JM, Moore HM, Giltnane J, Friedman LS, Chow Maneval E, Chan I, Jhaveri K. The oral selective estrogen receptor degrader GDC-0810 (ARN-810) in postmenopausal women with hormone receptor-positive HER2-negative (HR + /HER2 -) advanced/metastatic breast cancer. Breast Cancer Res Treat. 2023 Jan;197(2):319-331. doi: 10.1007/s10549-022-06797-9. Epub 2022 Nov 19. PMID 36401732

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9 | Phase IIa - Cohort A1 | Phase IIa - Cohort A2 | Phase IIa - Cohort B1 | Phase IIa - Cohort B2 | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
Started | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3 | 19 | 10 | 53 | 19 | 4 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3 | 19 | 10 | 53 | 19 | 4 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 4 | 3 | 6 | 4 | 6 | 5 | 3 | 3 | 18 | 8 | 46 | 18 | 4 | 6
Not completed — Study Termination | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9 | Phase IIa - Cohort A1 | Phase IIa - Cohort A2 | Phase IIa - Cohort B1 | Phase IIa - Cohort B2 | Phase Ib - Cohort C1 | Phase Ib - Cohort D1 | Total
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3 | 19 | 10 | 53 | 19 | 4 | 6 | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (5.7) | 63.5 (9.6) | 60.8 (6.9) | 55.3 (8.5) | 69.3 (7.2) | 56.2 (12.8) | 50.5 (14.6) | 58.3 (3.5) | 64.7 (4.0) | 55.4 (12.2) | 63.4 (8.9) | 61.9 (9.3) | 62.6 (12.2) | 58.5 (13.1) | 41.7 (8.9) | 59.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3 | 19 | 10 | 53 | 19 | 4 | 6 | 152
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity was only collected from 151 participants
  Participants
    Asian | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 3 | 10
    Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
    White | 2 | 4 | 3 | 6 | 5 | 4 | 6 | 3 | 3 | 17 | 8 | 46 | 15 | 4 | 1 | 127
    Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 0 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Phase Ia: Maximum Tolerated Dose of GDC-0810 When Used as a Single Agent
Description: Maximum Tolerated Dose (MTD) is determined based on the number of Dose Limiting Toxicities (DLTs) experienced by the participants. DLTs were defined as any of the following adverse events (AEs) that are deemed by the investigator or the Sponsor to be related to study drug (toxicities will be attributed to single agent GDC-0810 unless they are clearly related to disease progression or can clearly be attributed to a cause other than GDC-0810 administration):
  * Any grade ≥ 3 non-hematologic toxicity (excluding alopecia)
  * Any grade ≥ 3 hematologic toxicity of > 7 days' duration
  * Any grade toxicity that leads to study drug interruption of > 7 days' duration
Time Frame: Day -7 through the first cycle (28 days) of treatment (35 days total)
Population: All participants that were enrolled in Phase Ia of the study.
Measure: Number; unit: milligram (mg)
Groups:
- Phase Ia - All Cohorts: GDC-0810 single agent was administered orally on a continuous daily dosing regimen
Arm/Group | Phase Ia - All Cohorts
Number analyzed (Participants) | 41
milligram (mg) | NA — The MTD could not be determined.

2. Primary Outcome: Phase Ia: RP2D of GDC-0810 When Used as a Single Agent
Description: The recommended Phase II dose (RP2D) was based on the overall safety/tolerability and pharmacokinetic profile of GDC-0810.
Time Frame: Day -7 through the first cycle (28 days) of treatment (35 days total)
Population: All participants that were enrolled in Phase Ia of the study.
Measure: Number; unit: milligram (mg)
Arm/Group | Phase Ia - All Cohorts
Number analyzed (Participants) | 41
milligram (mg) | 600

3. Primary Outcome: Phase IIa: Percentage of Participants With Confirmed Objective Tumor Response of GDC-0810 According to RECIST v1.1
Description: Objective response (OR) is defined as a complete response (CR) or partial response (PR) as determined by investigator assessment according to RECIST v1.1. OR was based on criteria related to changes in size of target lesions. CR was the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Screening and every 8 weeks from Cycle 1 Day 1 until Cycle 12, thereafter every 3 months until disease progression (up to 3 years)
Population: All participants that were enrolled in Phase IIa of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Phase IIa - Cohort A1 | Phase IIa - Cohort A2 | Phase IIa - Cohort B1 | Phase IIa - Cohort B2
Number analyzed (Participants) | 19 | 10 | 53 | 19
percentage of participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 7.5 | 0

4. Primary Outcome: Phase IIa: Percentage of Participants With Clinical Benefit Response of GDC-0810 According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Clinical Benefit Response (CBR) is defined as the percentage of participants achieving confirmed RECIST v1.1 defined CR, PR, and/or stable disease. CR was the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: as for outcome 3
Population: All participants that were enrolled in Phase IIa of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Phase IIa - Cohort A1 | Phase IIa - Cohort A2 | Phase IIa - Cohort B1 | Phase IIa - Cohort B2
Number analyzed (Participants) | 19 | 10 | 53 | 19
percentage of participants | 5.3 | 10.0 | 28.3 | 15.8

5. Primary Outcome: Phase Ib: RP2D of GDC-0810 When Used in Combination With Palbociclib and/or LHRH
Description: The RP2D of GDC-0810 When Used in Combination With Palbociclib and/or LHRH RP2D was not determined since the development of the GDC-0810 was discontinued before enrolling Cohort C2. The RP2D would have been based on the overall safety and PK/PD profile of GDC-0810 and palbociclib, and not necessarily the MTD.
Time Frame: first cycle (Days 1 to 28 of a 28-day schedule)
Population: All participants that were enrolled in Phase Ib of the study.
Measure: Number; unit: mg
Arm/Group | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
Number analyzed (Participants) | 4 | 6
mg | NA — Due to discontinuation of GDC-0810 development, data is limited and RP2D was not determined | NA — Due to discontinuation of GDC-0810 development, data is limited and RP2D was not determined

6. Secondary Outcome: All Phases: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Time Frame: up to 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9 | Phase IIa - Cohort A1 | Phase IIa - Cohort A2 | Phase IIa - Cohort B1 | Phase IIa - Cohort B2 | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3 | 19 | 10 | 53 | 19 | 4 | 6
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100

7. Secondary Outcome: Phase Ia: Maximum Plasma Concentration (Cmax) of GDC-0810 Single Agent and Its Glucuronide Metabolites
Description: Maximum Plasma Concentration (Cmax) has been calculated using PK samples collected after administration of a single dose (on Day -7) and also following once-daily multiple doses (at steady state on Day 29) of GDC-0810.
Time Frame: Single Dose: Day-7 at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48 hours postdose; Multiple Doses: Day 29 (Cycle 2 Day 1) at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, hours postdose
Population: All participants that were enrolled in Phase Ia of the study and provided sufficient blood samples for analysis.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3
micrograms per milliliter (ug/mL)
  GDC-0810 (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 3
  GDC-0810 (Single Dose) | 2.29 (1.24) | 3.76 (0.599) | 9.4 (2.53) | 12.7 (5.36) | 22.2 (11.6) | 9.73 (4.5) | 15.9 (3.13) | 15.6 (4.97) | 10.1 (4.23)
  GDC-0810 (Multiple Doses): number analyzed (Participants) | 3 | 3 | 4 | 6 | 5 | 5 | 4 | 3 | 3
  GDC-0810 (Multiple Doses) | 2.59 (1.43) | 3.26 (1.11) | 9.08 (3.43) | 11.8 (6.61) | 25 (8.35) | 8.89 (3.96) | 18.4 (4.84) | 25.5 (9.3) | 13.9 (4.87)
  GDC-0810-N-Glucuronide (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 3
  GDC-0810-N-Glucuronide (Single Dose) | 0.0171 (0.021) | 0.0535 (0.015) | 0.177 (0.1) | 0.468 (0.388) | 0.691 (0.526) | 0.299 (0.171) | 1.38 (1.19) | 0.369 (0.338) | 0.153 (0.0421)
  GDC-0810-N-Glucuronide (Multiple Doses): number analyzed (Participants) | 3 | 3 | 4 | 6 | 5 | 5 | 4 | 3 | 3
  GDC-0810-N-Glucuronide (Multiple Doses) | 0.067 (0.055) | 0.061 (0.0271) | 0.184 (0.0832) | 0.416 (0.346) | 0.723 (0.338) | 0.181 (0.0846) | 0.74 (0.327) | 1.17 (0.893) | 0.308 (0.148)
  GDC-0810-Acyl-Glucuronide (Single Dose): number analyzed (Participants) | 0 | 0 | 4 | 2 | 6 | 6 | 4 | 3 | 3
  GDC-0810-Acyl-Glucuronide (Single Dose) |  |  | 1.46 (0.997) | 3 (0.827) | 2.26 (1.24) | 1.35 (0.876) | 7.02 (8.19) | 1.29 (0.617) | 1.36 (0.421)
  GDC-0810-Acyl-Glucuronide (Multiple Doses): number analyzed (Participants) | 0 | 0 | 4 | 2 | 5 | 5 | 4 | 3 | 3
  GDC-0810-Acyl-Glucuronide (Multiple Doses) |  |  | 1.89 (1.34) | 3.64 (2.96) | 3.16 (1.2) | 0.993 (0.435) | 3.37 (2.34) | 4.62 (2.19) | 2.82 (1.43)

8. Secondary Outcome: Phase Ia: Time to Maximum Concentration (Tmax) of GDC-0810 Single Agent and Its Glucuronide Metabolites
Description: Time to Maximum Concentration (Tmax) has been calculated using PK samples collected after administration of a single dose (on Day -7) and also following once-daily multiple doses (at steady state on Day 29) of GDC-0810.
Time Frame: as for outcome 7
Population: All participants that were enrolled in Phase Ia of the study and provided sufficient blood samples for analysis.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3
hour (hr)
  GDC-0810 (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 2 | 3
  GDC-0810 (Single Dose) | 1.5 [1.5 to 2] | 1.71 [1.45 to 2] | 2 [1 to 3] | 2.99 [1.25 to 4] | 3.01 [1.5 to 6] | 1.48 [0.217 to 3.03] | 3.04 [2.17 to 4] | 2 [2 to 4.07] | 1.88 [1 to 3]
  GDC-0810 (Multiple Doses): number analyzed (Participants) | 3 | 3 | 4 | 6 | 5 | 5 | 4 | 3 | 3
  GDC-0810 (Multiple Doses) | 1.47 [0.95 to 2] | 0.9 [0.45 to 1] | 1.55 [1.07 to 1.68] | 2.48 [1.93 to 6.45] | 2.95 [1.95 to 4.03] | 1.65 [0.917 to 3.07] | 1.59 [1.08 to 1.92] | 2.93 [1.53 to 6.3] | 2.05 [1.47 to 2.42]
  GDC-0810-N-Glucuronide (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 3
  GDC-0810-N-Glucuronide (Single Dose) | 0.5 [0.5 to 1.5] | 1.95 [1.5 to 2] | 2 [1.52 to 3] | 2.85 [2 to 4] | 3.51 [1.5 to 6.07] | 1.72 [0.217 to 3.03] | 3.54 [3 to 4] | 3 [2 to 4.07] | 1.88 [1 to 3]
  GDC-0810-N-Glucuronide (Multiple Doses): number analyzed (Participants) | 3 | 3 | 4 | 6 | 5 | 5 | 4 | 3 | 3
  GDC-0810-N-Glucuronide (Multiple Doses) | 2 [0 to 2.05] | 1 [0.9 to 1.48] | 1.64 [1.52 to 2.08] | 3.49 [1.93 to 4.45] | 2.95 [1.95 to 4.03] | 1.65 [0.917 to 3.07] | 2.27 [1.08 to 3.03] | 2.93 [1.53 to 6.3] | 2.05 [1.47 to 3.37]
  GDC-0810-Acyl-Glucuronide (Single Dose): number analyzed (Participants) | 0 | 0 | 4 | 2 | 6 | 6 | 4 | 3 | 3
  GDC-0810-Acyl-Glucuronide (Single Dose) |  |  | 2 [1.52 to 3] | 2.85 [2.72 to 2.98] | 3.51 [2 to 6.07] | 1.98 [0.717 to 3.03] | 3.54 [3 to 4] | 3 [2 to 4.07] | 2.98 [1 to 3]
  GDC-0810-Acyl-Glucuronide (Multiple Doses): number analyzed (Participants) | 0 | 0 | 4 | 2 | 5 | 5 | 4 | 3 | 3
  GDC-0810-Acyl-Glucuronide (Multiple Doses) |  |  | 1.84 [1.52 to 2.17] | 3.53 [3.07 to 4] | 2.95 [1.95 to 4.03] | 1.65 [0.917 to 3.07] | 2.27 [1.08 to 3.03] | 2.93 [1.53 to 6.3] | 2.05 [2 to 3.37]

9. Secondary Outcome: Phase Ia: Area Under the Concentration-time Curves at 6 Hours (AUC0-6) of GDC-0810 Single Agent and Its Glucuronide Metabolites
Description: Area under the concentration-time curves from time 0 to 6 hours (AUC0-6) has been calculated using PK samples collected after administration of a single dose (on Day -7) and also following once-daily multiple doses (at steady state on Day 29) of GDC-0810.
Time Frame: Single Dose: Day-7 at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6 hours postdose; Multiple Doses: Day 29 (Cycle 2 Day 1) at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6 hours postdose
Population: All participants that were enrolled in Phase Ia of the study and provided sufficient blood samples for analysis.
Measure: Mean (Standard Deviation); unit: hr*ug/mL
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3
hr*ug/mL
  GDC-0810 (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 3
  GDC-0810 (Single Dose) | 3.18 (1.65) | 6.78 (1.19) | 23.7 (11.3) | 34.3 (14.4) | 58.2 (28.9) | 18.8 (7.38) | 51.1 (18) | 48.3 (28.4) | 22.1 (5.43)
  GDC-0810 (Multiple Doses): number analyzed (Participants) | 3 | 3 | 4 | 6 | 5 | 5 | 3 | 3 | 3
  GDC-0810 (Multiple Doses) | 4.83 (2.3) | 6.19 (2.18) | 18.8 (4.76) | 41.1 (27.5) | 74.9 (30.1) | 19.3 (7.01) | 65.7 (20.6) | 70.5 (22) | 43 (26)
  GDC-0810-N-Glucuronide (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 3
  GDC-0810-N-Glucuronide (Single Dose) | 0.0401 (0.0197) | 0.116 (0.0729) | 0.321 (0.149) | 1.16 (0.815) | 1.36 (0.917) | 0.486 (0.36) | 3.81 (4.15) | 0.938 (0.983) | 0.29 (0.0295)
  GDC-0810-N-Glucuronide (Multiple Doses): number analyzed (Participants) | 3 | 3 | 4 | 6 | 5 | 5 | 3 | 3 | 3
  GDC-0810-N-Glucuronide (Multiple Doses) | 0.105 (0.0724) | 0.103 (0.0335) | 0.321 (0.105) | 1.37 (1.21) | 1.83 (1.01) | 0.409 (0.23) | 2.63 (1.01) | 2.08 (1.15) | 0.974 (0.605)
  GDC-0810-Acyl-Glucuronide (Single Dose): number analyzed (Participants) | 0 | 0 | 4 | 2 | 6 | 6 | 4 | 3 | 3
  GDC-0810-Acyl-Glucuronide (Single Dose) |  |  | 3.18 (1.77) | 8.25 (4.54) | 5.29 (2.71) | 2.76 (2.23) | 21.1 (26.9) | 3.99 (2.29) | 3.27 (1.03)
  GDC-0810-Acyl-Glucuronide (Multiple Doses): number analyzed (Participants) | 0 | 0 | 4 | 2 | 5 | 5 | 3 | 3 | 3
  GDC-0810-Acyl-Glucuronide (Multiple Doses) |  |  | 3.72 (1.91) | 13 (11.1) | 8.25 (3.47) | 2.03 (0.669) | 14 (11.1) | 10.2 (3.61) | 8.45 (5.79)

10. Secondary Outcome: Phase Ia: Area Under the Concentration-time Curves at 24 Hours (AUC0-24) of GDC-0810 Single Agent and Its Glucuronide Metabolites
Description: Area under the concentration-time curves from time 0 to 24 hours (AUC0-24) has been calculated using PK samples collected after administration of a single dose (on Day -7) and also following once-daily multiple doses (at steady state on Day 29) of GDC-0810.
Time Frame: Single Dose: Day-7 at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours postdose; Multiple Doses: Day 29 (Cycle 2 Day 1) at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24 hours postdose
Population: All participants that were enrolled in Phase Ia of the study and provided sufficient blood samples for analysis.
Measure: Mean (Standard Deviation); unit: hr*ug/mL
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9
Number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 6 | 3 | 3
hr*ug/mL
  GDC-0810 (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 3
  GDC-0810 (Single Dose) | 3.58 (1.75) | 8.81 (2.52) | 28.5 (15.6) | 44.7 (19.5) | 101 (49.9) | 41.2 (15.9) | 61.8 (25.5) | 95.1 (76.4) | 47.7 (11.4)
  GDC-0810 (Multiple Doses): number analyzed (Participants) | 2 | 3 | 4 | 6 | 5 | 5 | 3 | 2 | 3
  GDC-0810 (Multiple Doses) | 5.34 (2.99) | 7.36 (1.32) | 22.8 (6.14) | 66.9 (46.8) | 102 (35.9) | 44.2 (14.5) | 80.4 (26.8) | 75.2 (15.4) | 109 (73.3)
  GDC-0810-N-Glucuronide (Single Dose): number analyzed (Participants) | 3 | 4 | 4 | 6 | 6 | 6 | 4 | 3 | 3
  GDC-0810-N-Glucuronide (Single Dose) | 0.13 (0.0197) | 0.224 (0.109) | 0.413 (0.152) | 1.54 (1.08) | 2.08 (1.02) | 1.07 (0.786) | 5.67 (7.17) | 1.83 (2.04) | 0.649 (0.055)
  GDC-0810-N-Glucuronide (Multiple Doses): number analyzed (Participants) | 2 | 3 | 4 | 6 | 5 | 5 | 3 | 2 | 3
  GDC-0810-N-Glucuronide (Multiple Doses) | 0.13 (0.0141) | 0.132 (0.0253) | 0.413 (0.121) | 2.63 (2.21) | 2.64 (1.4) | 1.09 (0.594) | 3.72 (1.81) | 2.35 (1.57) | 2.66 (1.58)
  GDC-0810-Acyl-Glucuronide (Single Dose): number analyzed (Participants) | 0 | 0 | 4 | 2 | 6 | 6 | 4 | 3 | 3
  GDC-0810-Acyl-Glucuronide (Single Dose) |  |  | 3.76 (2.13) | 11.4 (7.43) | 8.59 (3.82) | 6.03 (4.89) | 30.6 (44) | 7.64 (5.51) | 7.1 (1.96)
  GDC-0810-Acyl-Glucuronide (Multiple Doses): number analyzed (Participants) | 0 | 0 | 4 | 6 | 6 | 5 | 3 | 2 | 3
  GDC-0810-Acyl-Glucuronide (Multiple Doses) |  |  | 4.42 (2.27) | 21.8 (21.2) | 10.4 (4.07) | 4.61 (1.34) | 18.1 (16.3) | 12 (5.44) | 20.8 (14.9)

11. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-Inf)
Description: Area under the concentration-time curve from time 0-infinity (AUC0-inf) has been calculated using PK samples collected after administration of a single dose (on Day -7) of GDC-0810.
Time Frame: Day-7 at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, and 48 hours postdose
Population: All participants that were enrolled in Phase Ia of the study, provided sufficient blood samples for analysis and received once daily dosing.
Measure: Mean (Standard Deviation); unit: hr*ug/ml
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 6 | 0 | 4 | 3 | 0
hr*ug/ml | 5.3 (1.96) | 10 (2.8) | 30.8 (16.3) | 40.5 (11.3) | 114 (57.4) |  | 65.7 (28) | 101 (78.5) |

12. Secondary Outcome: Phase Ia: Plasma Half-life (t1/2) of GDC-0810 Single Agent
Description: Half-life (t1/2) was calculated after single dose administration and not at steady state.
Time Frame: Day -7 at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48 hours postdose
Population: All participants that were enrolled in Phase Ia of the study and provided sufficient blood samples for analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 6 | 6 | 4 | 3 | 3
hr | 40.7 (3.47) | 15.2 (2.35) | 24.1 (17.3) | 9.58 (3.41) | 7.91 (2.67) | NA (NA) — t1/2 can be estimated only when the PK sample collection following a dose is long enough to characterize the elimination phase. With twice-daily dosing (BID), the PK samples were collected for only up to 6 hours following a dose (after which the patients received their next dose), which is not sufficient to estimate t1/2. Therefore, t1/2 was not reported for BID cohorts. | 10.1 (1.59) | 7.09 (3.23) | NA (NA) — t1/2 can be estimated only when the PK sample collection following a dose is long enough to characterize the elimination phase. With twice-daily dosing (BID), the PK samples were collected for only up to 6 hours following a dose (after which the patients received their next dose), which is not sufficient to estimate t1/2. Therefore, t1/2 was not reported for BID cohorts.

13. Secondary Outcome: Phase Ia: Apparent Clearance (Cl/F)
Description: Apparent Clearance (CL/F) was estimated using PK samples collected following administration of a single dose (on Day -7) of GDC-0810
Time Frame: Day -7 at 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 48 hours postdose
Population: All participants that were enrolled in Phase Ia of the study and provided sufficient blood samples for analysis.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 6 | 6 | 4 | 3 | 3
L/hr | 20.4 (6.43) | 21 (4.94) | 15.1 (5.56) | 15.7 (4.13) | 8.21 (8.38) | NA (NA) — CL/F can be estimated only when the PK sample collection following a dose is long enough to characterize the elimination phase. With BID dosing, the PK samples were collected for only up to 6 hours before the patient received their next dose, which is not sufficient to estimated CL/F. Therefore, CL/F was not reported for BID cohorts. | 15.1 (9.45) | 11.1 (6.23) | NA (NA) — CL/F can be estimated only when the PK sample collection following a dose is long enough to characterize the elimination phase. With BID dosing, the PK samples were collected for only up to 6 hours before the patient received their next dose, which is not sufficient to estimated CL/F. Therefore, CL/F was not reported for BID cohorts.

14. Secondary Outcome: Phase IIa: Effect of GDC-0810 Single Agent on Ventricular Repolarization as Measured by Corrected QT Intervals (QTc) Using Fridericia's Formula
Description: The corrected QT interval (QTc) was calculated using Fridericia's formula from electrocardiogram (ECG) data. Changes in ECG intervals from baseline were calculated. Triplicate ECG measurements were collected throughout the study. The averaged triplicate ECG measurements were used for analysis.
Time Frame: Screening; on Cycle 2 Day 1 predose and at 1, 2, 3, 4, and 6 hours postdose; Cycle 3 Day 1 predose, and at 1, 3, and 6 hours post dose
Population: All participants enrolled in Phase IIa of the study and with post baseline ECG measurements
Measure: Number; unit: percentage of participants
Arm/Group | Phase IIa - Cohort A1 | Phase IIa - Cohort A2 | Phase IIa - Cohort B1 | Phase IIa - Cohort B2
Number analyzed (Participants) | 13 | 3 | 34 | 11
percentage of participants
  ≤ 450 milliseconds (msec) | 100 | 66.7 | 91.2 | 100
  >450 and ≤480 msec | 0 | 33.3 | 8.8 | 0
  Increase from baseline ≤30 msec: number analyzed (Participants) | 13 | 3 | 33 | 11
  Increase from baseline ≤30 msec | 100 | 100 | 93.9 | 100
  Increase from baseline >30 and ≤60 msec: number analyzed (Participants) | 13 | 3 | 33 | 11
  Increase from baseline >30 and ≤60 msec | 0 | 0 | 6.1 | 0

15. Secondary Outcome: Phase Ib: Cmax of GDC-0810 in Combination With Palbociclib and/or an LHRH Agonist
Description: Cmax has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: C1: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 8; D1: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: All participants that were enrolled in Phase Ib of the study and provided sufficient samples for analysis.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
Number analyzed (Participants) | 4 | 3
ug/ml
  Cycle 1 Day 1 (C1D1) | 10.2 (2.98) | 8.96 (1.87)
  Cycle 1 Day 8 (C1D8): number analyzed (Participants) | 4 | 0
  Cycle 1 Day 8 (C1D8) | 9.95 (5.85) |
  Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 0 | 2
  Cycle 2 Day 1 (C2D1) |  | 9.62 (0.0354)

16. Secondary Outcome: Phase Ib: Tmax of GDC-0810 in Combination With Palbociclib and/or an LHRH Agonist
Description: Tmax has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: as for outcome 15
Population: All participants that were enrolled in Phase Ib of the study and provided sufficient samples for analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
Number analyzed (Participants) | 4 | 3
hr
  C1D1 | 2 [1 to 6] | 3 [2 to 4]
  C1D8: number analyzed (Participants) | 4 | 0
  C1D8 | 2.5 [1 to 6] |
  C2D1: number analyzed (Participants) | 0 | 3
  C2D1 |  | 3 [3 to 3]

17. Secondary Outcome: Phase Ib: AUC0-6 of GDC-0810 in Combination With Palbociclib and/or an LHRH Agonist
Description: AUC0-6 has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: as for outcome 15
Population: All participants that were enrolled in Phase Ib of the study.
Measure: Mean (Standard Deviation); unit: hr*ug/ml
Arm/Group | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
Number analyzed (Participants) | 4 | 3
hr*ug/ml
  C1D1 | 18.9 (9.19) | 33.6 (7.91)
  C1D8: number analyzed (Participants) | 4 | 0
  C1D8 | 18.2 (10.4) |
  C2D1: number analyzed (Participants) | 0 | 2
  C2D1 |  | 38.8 (3.53)

18. Secondary Outcome: Phase Ib: t/2 of GDC-0810 in Combination With Palbociclib and/or an LHRH Agonist
Description: Half-life (t1/2) can be estimated only when the PK sample collection following a dose is long enough to characterize the elimination phase. The PK samples in these cohorts were only collected up to 6 hours following the dose, hence, t1/2 could not be estimated.
Time Frame: as for outcome 15
Population: No data from any participants could be used for analysis.
Arm/Group | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Phase Ib: Cmax of Palbociclib in Combination With GDC-0810 and/or an LHRH Agonist
Description: Cmax has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: All participants that were enrolled in Phase Ib of the study, Cohort C1 and provided sufficient samples for analysis.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Phase Ib - Cohort C1
Number analyzed (Participants) | 4
ug/ml
  C1D1: number analyzed (Participants) | 3
  C1D1 | 54.8 (9.04)
  C1D8 | 97.8 (27.1)

20. Secondary Outcome: Phase Ib: Tmax of Palbociclib in Combination With GDC-0810 and/or an LHRH Agonist
Description: Tmax has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: All participants that were enrolled in Phase Ib of the study, Cohort C1 and provided sufficient samples for analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Phase Ib - Cohort C1
Number analyzed (Participants) | 4
hr
  C1D1: number analyzed (Participants) | 3
  C1D1 | 4 [3 to 6]
  C1D8 | 6 [0 to 6]

21. Secondary Outcome: Phase Ib: AUC0-6 of Palbociclib in Combination With GDC-0810 and/or an LHRH Agonist
Description: AUC0-6 has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: All participants that were enrolled in Phase Ib of the study, Cohort C1 and provided sufficient samples for analysis.
Measure: Mean (Standard Deviation); unit: hr*ug/ml
Arm/Group | Phase Ib - Cohort C1
Number analyzed (Participants) | 4
hr*ug/ml
  C1D1: number analyzed (Participants) | 3
  C1D1 | 200 (41.4)
  C1D8 | 464 (106)

22. Secondary Outcome: Phase Ib: t/2 of Palbociclib in Combination With GDC-0810 and/or an LHRH Agonist
Description: as for outcome 18
Time Frame: Cohort C1: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 1 Day 8
Population: No data from any participants could be used for analysis.
Arm/Group | Phase Ib - Cohort C1
Number analyzed (Participants) | 0

23. Secondary Outcome: Phase Ib: Cmax of LHRH Agonist in Combination With GDC-0810 and/or Palbociclib
Description: Cmax has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: All participants that were enrolled in Phase Ib of the study, Cohort D1 and provided sufficient samples for analysis.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Phase Ib - Cohort D1
Number analyzed (Participants) | 3
ug/ml
  C1D1 | 39.6 (9.85)
  C2D1: number analyzed (Participants) | 1
  C2D1 | 32.4 (NA) — The Standard Deviation is not applicable as the results data are reported for 1 participant only.

24. Secondary Outcome: Phase Ib: Tmax of LHRH Agonist in Combination With GDC-0810 and/or Palbociclib
Description: Tmax has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: All participants that were enrolled in Phase Ib of the study, Cohort D1 and provided sufficient samples for analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Phase Ib - Cohort D1
Number analyzed (Participants) | 3
hr
  C1D1 | 3 [2 to 6]
  C1D8: number analyzed (Participants) | 1
  C1D8 | 3 [NA to NA] — The Range is not applicable as the results data are reported for 1 participant only.

25. Secondary Outcome: Phase Ib: AUC0-6 of LHRH Agonist in Combination With GDC-0810 and/or an Palbociclib
Description: AUC0-6 has been calculated using PK samples collected after GDC-0810 administration.
Time Frame: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: All participants that were enrolled in Phase Ib of the study, Cohort D1 and provided sufficient samples for analysis.
Measure: Mean (Standard Deviation); unit: hr*ug/ml
Arm/Group | Phase Ib - Cohort D1
Number analyzed (Participants) | 3
hr*ug/ml
  C1D1 | 118 (76.4)
  C2D1: number analyzed (Participants) | 1
  C2D1 | 106 (NA) — The Standard Deviation is not applicable as the results data are reported for 1 participant only.

26. Secondary Outcome: Phase Ib: t/2 of LHRH Agonist in Combination With GDC-0810 and/or Palbociclib
Description: as for outcome 18
Time Frame: Cohort D1: Predose and at 1, 2, 3, 4, and 6 hours postdose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: No data from any participants could be used for analysis.
Arm/Group | Phase Ib - Cohort D1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Phase Ia - Cohort 1 | Phase Ia - Cohort 2 | Phase Ia - Cohort 3 | Phase Ia - Cohort 4 | Phase Ia - Cohort 5 | Phase Ia - Cohort 6 | Phase Ia - Cohort 7 | Phase Ia - Cohort 8 | Phase Ia - Cohort 9 | Phase IIa - Cohort A1 | Phase IIa - Cohort A2 | Phase IIa - Cohort B1 | Phase IIa - Cohort B2 | Phase Ib - Cohort C1 | Phase Ib - Cohort D1
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/4 | 0/4 | 1/6 | 2/6 | 0/6 | 1/6 | 0/3 | 0/3 | 0/19 | 0/10 | 3/53 | 0/19 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 1/4 | 1/6 | 3/6 | 4/6 | 1/6 | 1/3 | 0/3 | 4/19 | 1/10 | 11/53 | 1/19 | 1/4 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 4/4 | 6/6 | 6/6 | 6/6 | 6/6 | 3/3 | 3/3 | 18/19 | 10/10 | 51/53 | 19/19 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ia - Cohort 1 (N=3) | Phase Ia - Cohort 2 (N=4) | Phase Ia - Cohort 3 (N=4) | Phase Ia - Cohort 4 (N=6) | Phase Ia - Cohort 5 (N=6) | Phase Ia - Cohort 6 (N=6) | Phase Ia - Cohort 7 (N=6) | Phase Ia - Cohort 8 (N=3) | Phase Ia - Cohort 9 (N=3) | Phase IIa - Cohort A1 (N=19) | Phase IIa - Cohort A2 (N=10) | Phase IIa - Cohort B1 (N=53) | Phase IIa - Cohort B2 (N=19) | Phase Ib - Cohort C1 (N=4) | Phase Ib - Cohort D1 (N=6)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC HAEMORRHAGE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ia - Cohort 1 (N=3) | Phase Ia - Cohort 2 (N=4) | Phase Ia - Cohort 3 (N=4) | Phase Ia - Cohort 4 (N=6) | Phase Ia - Cohort 5 (N=6) | Phase Ia - Cohort 6 (N=6) | Phase Ia - Cohort 7 (N=6) | Phase Ia - Cohort 8 (N=3) | Phase Ia - Cohort 9 (N=3) | Phase IIa - Cohort A1 (N=19) | Phase IIa - Cohort A2 (N=10) | Phase IIa - Cohort B1 (N=53) | Phase IIa - Cohort B2 (N=19) | Phase Ib - Cohort C1 (N=4) | Phase Ib - Cohort D1 (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (3) | 3 (3) | 4 (13) | 1 (2) | 1 (3) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 6 (6) | 4 (8) | 2 (2) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BLEPHARITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 10 (11) | 1 (3) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 6 (11) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 4 (7) | 2 (2) | 2 (2) | 2 (5) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 16 (21) | 4 (4) | 0 (0) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (2) | 4 (11) | 4 (6) | 6 (22) | 4 (12) | 6 (21) | 3 (7) | 3 (6) | 10 (16) | 5 (11) | 28 (66) | 11 (30) | 2 (2) | 6 (13)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 6 (8) | 2 (2) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 6 (6) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 3 (3)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
ERUCTATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 13 (14) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 9 (10) | 3 (5) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (4) | 6 (11) | 2 (3) | 4 (4) | 6 (15) | 2 (2) | 2 (7) | 8 (9) | 6 (6) | 24 (32) | 9 (10) | 3 (6) | 4 (8)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 1 (3) | 1 (3) | 4 (15) | 3 (5) | 2 (4) | 7 (11) | 4 (5) | 14 (22) | 2 (2) | 0 (0) | 3 (5)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
FATIGUE (General disorders) | 1 (2) | 1 (2) | 3 (3) | 5 (7) | 5 (6) | 2 (2) | 6 (12) | 2 (3) | 3 (7) | 8 (9) | 2 (3) | 27 (29) | 7 (7) | 2 (2) | 3 (3)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
IMPAIRED HEALING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SWELLING FACE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TENDERNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (2) | 1 (1) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (1) | 0 (0) | 3 (8) | 3 (5) | 3 (4) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (1) | 0 (0) | 4 (6) | 3 (4) | 4 (7) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD URIC ACID INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
LIVER FUNCTION TEST INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 2 (3) | 2 (10) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (6) | 6 (6) | 3 (3) | 9 (9) | 2 (2) | 1 (1) | 4 (4)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 2 (3) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 2 (2) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (3) | 4 (5) | 0 (0) | 14 (18) | 0 (0) | 1 (1) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 13 (15) | 4 (4) | 2 (2) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 1 (1) | 1 (1) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (5) | 2 (2) | 0 (0) | 2 (2)
NECK MASS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (12) | 1 (1) | 1 (1) | 2 (3)
HYPERSOMNIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
TASTE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
MOOD SWINGS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BREAST ATROPHY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRIAL THICKENING (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OEDEMA GENITAL (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 9 (9) | 0 (0) | 8 (9) | 4 (4) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 8 (11) | 5 (6) | 1 (4) | 1 (1)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAPULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (6) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 10 (11) | 9 (9) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
PALLOR (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXTERNAL EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IDIOPATHIC ORBITAL INFLAMMATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHOTOPSIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECES SOFT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVAL SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIP SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL MUCOSAL ERUPTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACIAL PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROUP INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HELICOBACTER INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AMYLASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
BLOOD CHLORIDE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CRYSTAL URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLUCOSE URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIGH DENSITY LIPOPROTEIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIGH DENSITY LIPOPROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NITRITE URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RED BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY CASTS PRESENT (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERPROTEINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IRRITABILITY (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MOOD ALTERED (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL DISORDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPAREUNIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LICHEN SCLEROSUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MACULE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MADAROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT01823835/Prot_SAP_000.pdf